CLINICAL TRIAL: NCT06782347
Title: Activating SilverSneakers Benefits for Seniors With Osteoarthritis: Proactive Versus Usual Care
Brief Title: Activating SilverSneakers Benefits for Seniors With Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Humana Healthcare Research (Unknown); Kaiser Permanente (Other); Global Healthy Living Foundation (Other); Patient-Centered Outcomes Research Institute (Other); CVS Healthspire Life Sciences Solutions (Unknown); Tivity Health (Unknown)
Responsible Party: Principal Investigator, Liza Rovniak, Associate Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BPS-2022C3-30497
Record Dates: First submitted 2024-06-25; First posted 2025-01-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis; Physical Inactivity
MeSH Terms: conditions — Osteoarthritis; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Care (Other): The Proactive Care condition will consist of one mailing to alert older adults to the existence of their SilverSneakers benefit, followed by two action-planning phone calls to prompt activation and use of the SilverSneakers exercise benefit. The action-planning calls will guide older adults through an action plan to enroll in SilverSneakers, and choose convenient joint-friendly SilverSneakers exercise options appropriate for their fitness level. Exercise options are available both in-person and online. Older adults will also be given the option to have an information sheet about SilverSneakers sent to their primary care providers to encourage further discussion about SilverSneakers.
  Interventions: Behavioral: Proactive Care
- Usual Care (No Intervention): The Usual Care condition will include the standard information provided to Medicare Advantage beneficiaries about SilverSneakers.

INTERVENTIONS:
Behavioral: Proactive Care — The proactive care intervention was designed to be similar to proactive care approaches used successfully in the tobacco control area. These proactive care procedures have not yet been adequately evaluated in the exercise promotion area.
  Arms: Proactive Care

SUMMARY:
The aim of this pragmatic randomized controlled trial is to test the effects of a brief proactive care intervention involving mailed material and two phone calls on: (1) increasing participation in SilverSneakers exercise programs among older adults with osteoarthritis; (2) improving physical, social and psychological outcomes identified as important to older adults with osteoarthritis; and (3) reducing costly osteoarthritis-related health service use. Approximately 1,454 older adults with osteoarthritis who have SilverSneakers access through their Medicare Advantage plan, but no prior SilverSneakers use, will be recruited to participate across the United States. Key outcome measures will be assessed over a two-year follow-up period.

DETAILED DESCRIPTION:
Exercise is an evidence-based strategy for managing osteoarthritis, but fewer than 15% of older adults exercise regularly. Lack of access to affordable fitness facilities and resources is often identified by older adults as a key barrier to regular exercise. However, more than half of U.S. older adults are enrolled in Medicare Advantage plans which include no-cost access to SilverSneakers or other similar exercise benefits. SilverSneakers benefits provide access to more than 15,000 fitness centers/gyms nationwide, and access to online- and in-person exercise classes taught at multiple fitness levels-all at no extra cost for older adults who are enrolled in participating Medicare Advantage plans. Remarkably, fewer than one-third of older adults use their insurance-covered SilverSneakers exercise benefits; with most unaware that they have access to these exercise benefits.

The investigators plan to conduct a pragmatic randomized controlled trial to compare the effects of Proactive Care, involving mailed material and phone calls plus a faxed information sheet for older adults' primary care providers, relative to Usual Care, involving the standard insurance-benefit information packet provided to older adults, on: (1) increasing participation in SilverSneakers exercise programs; (2) improving physical, social, and psychological outcomes identified as important to patients; and (3) reducing osteoarthritis-related health service use. Approximately 1,454 older adults who are enrolled in a Medicare Advantage plan at Humana and have no prior SilverSneakers use will be recruited across the United States. Participants will be followed over a 2-year period for key outcomes, with assessments conducted at baseline, 6, 12, and 24 months. Outcome measures will be obtained from Humana health claims databases and from self-report surveys.

The investigators hypothesize that, relative to the Usual Care group, the Proactive Care group will result in: (1) a greater proportion of participants who enroll in, and use SilverSneakers at least once; (2) a greater proportion of participants who use SilverSneakers at least one time per month at 2-year follow-up; and (3) greater mean improvements in physical functioning between baseline and 2-year follow-up. If these hypotheses are supported, and if proactive care procedures improve exercise participation and health outcomes and reduce costly health-service use, it could lead health insurers to adopt proactive care procedures more widely. Using proactive care procedures on a wider scale holds potential to help millions of older adults with osteoarthritis to access their insurance-covered exercise benefits, and improve the quality of their daily lives. Patient-, primary care-, community- and policy-level stakeholder partners will provide input throughout the project period to ensure the design, delivery and dissemination of proactive care procedures are patient-centered and incorporate diverse stakeholder perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and older.
* ICD-9 or ICD-10 code for hip, knee, or general osteoarthritis.
* Positive response to a standardized question from the Medical Expenditure Panel Survey that asks if patient was diagnosed with osteoarthritis/arthritis and self-report confirmation of hip and/or knee pain due to their osteoarthritis/arthritis.
* Continuous enrollment for at least one year in a Humana Medicare Advantage plan which provides free SilverSneakers access and both medical and prescription drug coverage.
* Not currently or previously enrolled in SilverSneakers.
* Speak English or Spanish.
* Physical/mental capacity to provide informed consent, based on not having an ICD-9 or ICD-10 code for dementia and being able to answer three questions to verify comprehension of the informed consent form.

Exclusion Criteria:

* Another person in the same household is enrolling/enrolled in the study (to prevent treatment contamination, only one participant per household can participate).
* Medicare/Medicaid dual enrollment due to limited data accessibility for this group.
* Receiving hospice care or under long-term institutional care (Part C) due to limited data accessibility for this group.
* Receiving care from a provider credentialed through a delegated arrangement (i.e., delegated provider), due to limited data accessibility for this group.
* Lack of a valid mailing address in the Humana medical claims databases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1454 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Physical Function (subscale) | Administered at baseline and at 6-, 12-, and 24-month follow-up; reported score for the primary outcome is the change between baseline and 24-month follow-up.
  This measure is a subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); items measure ability to perform activities of daily living. Each item is scored on a 5-point Likert scale ranging from None (0) to Extreme (4). The scores are summed, with a possible score range of 0 to 68 for the Physical Function subscale. Higher scores indicate worse functional limitations.
SilverSneakers Activation | Obtained from Humana health claims databases at baseline and at 6-, 12-, and 24-month follow-up; the number of participants who enrolled in SilverSneakers and used the benefit is calculated as a cumulative total across all assessment points.
  Number of participants who enrolled in SilverSneakers and used their SilverSneakers benefit at least one time.
SilverSneakers Long-Term Participation Rate | Obtained from Humana health claims databases at 12- and 24-month follow-up; primary outcome measured at 24-month follow-up.
  Of those participants who enrolled in SilverSneakers and used their SilverSneakers benefit at least once, the number who are still using their SilverSneakers benefit ≥1 time/month at 24-month follow-up.

SECONDARY OUTCOMES:
SilverSneakers Usage Frequency | Obtained from Humana health claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Number of times per month participant used their SilverSneakers benefit.
SilverSneakers Interaction Mode | Obtained from Humana health claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  The interaction mode (e.g., in-person, online) of participants' SilverSneakers exercise activities.
Moderate-to-Vigorous Physical Activity and Strength Training | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Three questions from the National Health Interview Survey will assess the proportion of participants meeting national physical activity guidelines. Participants will be asked how many times per week they do leisure-time vigorous activities, light or moderate activities, and strength training. Scores range from 0 to 7 times per week with a higher score (more times per week) indicating better adherence to physical activity guidelines.
Pain (subscale) | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  This measure is a subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); items measure hip and knee pain while in motion and at rest. Each item is scored on a 5-point Likert scale ranging from None (0) to Extreme (4). The scores are summed, with a possible score range of 0 to 20 for the Pain subscale. Higher scores indicate worse pain.
Fatigue | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-short form. Each item is scored on a 5-point Likert scale ranging from Never (1) to Always (5). The scores are summed, with a possible score range of 7 to 35. Higher scores indicate greater fatigue.
Depression | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-short form. Each item is scored on a 5-point Likert scale ranging from Never (1) to Always (5). The scores are summed, with a possible score range of 8 to 40. Higher scores indicate greater severity of depression.
Loneliness | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Assessed by UCLA Brief Loneliness Scale. Each item is scored on a 3-point Likert scale ranging from Hardly Ever (1) to Often (3). The scores are summed, with a possible score range of 3 to 9. Higher scores indicate greater loneliness.
Satisfaction with Participation in Discretionary Social Activities | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS)-short form. Each item is scored on a 5-point Likert scale ranging from Not at All (1) to Very Much (5). The scores are summed, with a possible score range of 7 to 35. Higher scores indicate greater satisfaction with participation in discretionary social activities.
Social Networks | Administered at baseline and at 6-, 12-, and 24-month follow-up.
  Assessed by Berkman-Syme Social Network Index; items measure different components of social networks including marital status, number of close friends and relatives, membership in community/recreational organizations, and participation in religious services. Scores are summed across the different types of social network connections and range from 1 to 4. Higher scores indicate greater social connectedness.
Spoke to Primary Care Provider about SilverSneakers | Administered at 24-month follow-up.
  Reported question asking if participant ever spoke to primary care provider about SilverSneakers.
Number of Hip, Knee, or other Joint Replacement Surgeries | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Surgical procedures will be identified using Current Procedural Terminology (CPT) codes, Diagnosis-Related Group (DRG) codes, and International Classification of Diseases procedure codes (ICD Px).
Number of Arthroscopic Surgeries | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Surgical procedures will be identified using CPT, DRG, and ICD Px codes.
Number of Inpatient Hospital Visits and Emergency Department Visits | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Visits will be identified using bill types, revenue codes, and Place of Treatment (POT).
Number of Fall-Related Injuries Requiring Medical Care | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Fall-related injuries will be determined based on the presence of ICD Px injury codes for moderate to severe injuries (excluding non-fall-related injuries) and fall-related E-codes.
Number of Outpatient Primary Care, Specialist, and Physiotherapy Visits | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Visits will be identified using POT, revenue codes, CPT codes, Healthcare Common Procedure Coding System (HCPCS) codes and modifiers.
Number of Radiography/Imaging Procedures | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  These procedures will be identified using CPT codes, HCPCS codes, and revenue codes.
Number of Joint Injections (e.g., corticosteroids, hyaluronic acid) | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  These injections will be identified using CPT codes, HCPCS codes, and HCPCS J-codes.
Analgesic/NSAID Drug Use | Obtained from Humana medical claims databases at baseline and at 6-, 12-, and 24-month follow-up.
  Drug names (separately for branded vs. generic) will be obtained for prescription drugs.
Estimated Healthcare Costs | Health service and cost data will be obtained at baseline (the baseline measurement will include the 1-year period prior to proactive care delivery) and at 6-, 12-, and 24-month follow-up.
  Total estimated healthcare costs for the health service categories described above will be computed using health service data from the Humana health claims databases and cost data from the www.cms.gov cost sites.

CONTACTS AND LOCATIONS:
Overall Officials: Liza S. Rovniak, PhD, MPH, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No